CLINICAL TRIAL: NCT02480673
Title: EFFECT OF Salvia Hispanica L. ( CHIA ) IN THE BIOCHEMICAL METABOLIC SYNDROME COMPONENTS IN PATIENTS IN THE NATIONAL MEDICAL CENTER WEST OF THE MEXICAN SOCIAL SECURITY INSTITUTE
Brief Title: EFFECT OF Salvia Hispanica l. (CHIA) IN THE BIOCHEMICAL METABOLIC SYNDROME COMPONENTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Ana Elena Perez Verdin, Dr., Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R-2015-785-047
Record Dates: First submitted 2015-06-22; First posted 2015-06-24 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Metabolic Syndrome X
Keywords: Metabolic Syndrome X; Chia; Dyslipidemia
MeSH Terms: conditions — Metabolic Syndrome; Dyslipidemias | interventions — Salvia hispanica seed extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Free diet plus Chia (Experimental): This subjects will consume 1 cookie oatmeal with chia before breakfast and dinner for 90 days without changing their diet
  Interventions: Dietary Supplement: Chia
- Normocaloric diet plus chia (Experimental): This subjects will consume 1 cookie oatmeal with chia before breakfast and dinner for 90 days along with a normocaloric diet
  Interventions: Dietary Supplement: Chia; Behavioral: Normocaloric diet
- Normocaloric diet plus oatmeal (Active Comparator): This subjects will consume 1 cookie oatmeal before breakfast and dinner for 90 days along with a normocaloric diet
  Interventions: Dietary Supplement: Oatmeal; Behavioral: Normocaloric diet
- Normocaloric diet (Active Comparator): This subjects will only go under a normocaloric diet for 90 days
  Interventions: Behavioral: Normocaloric diet

INTERVENTIONS:
Dietary Supplement: Chia — The subject will eat 25 gr of chia in 2 oatmeal cookies at day
  Other Names: Salvia hispanica
  Arms: Free diet plus Chia; Normocaloric diet plus chia
Dietary Supplement: Oatmeal — The subject will eat 2 oatmeal cookies a day containing the exactly same quantity of oats in the oatmeal cookies with chia.
  Other Names: Oats
  Arms: Normocaloric diet plus oatmeal
Behavioral: Normocaloric diet — The healthy diet plan distribution will be 50% carbohydrate, 25 % protein, 35 % fat to less than 7 % saturated fat and less than 200 mg/d cholesterol and 20-30 g of fiber.
  Arms: Normocaloric diet; Normocaloric diet plus chia; Normocaloric diet plus oatmeal

SUMMARY:
The objective of this study is to evaluate the effect of the administration of 25 g of chia per day, for 90 days on the biochemical components of the metabolic syndrome in subjects with this condition

DETAILED DESCRIPTION:
The metabolic syndrome (MS) is a cardiovascular risk factor and is present in about 20-25% of the world's adult population. Individuals with this condition have twice the risk of cardiovascular disease and die from it, compared with those who do not and 5 times more likely to develop type 2 diabetes mellitus (DM2). For this reason, it is appropriate to develop better tools for prevention and management of MS, with more emphasis on lifestyle´s changes. Chia has been studied in the past 10 years due to its high concentration of omega-3 alpha-linolenic acid (ALA) and 6 linoleic acid (LA) showing beneficial effects in some components of MS in rodents and individuals. The addition of chia to the conventional treatment of MS for the modification of metabolic disorders provides us a tool for easy incorporation into daily life, inexpensive and accessible in our environment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metabolic syndrome according to Adult Treatment Panel - III criteria.
* Subject wishing to participate in the study by written consent.
* Instituto Mexicano del Seguro Social beneficiaries subject
* Subject who not requiring modification of medical treatment for MS in the recruitment period.

Exclusion Criteria:

* Chronic renal failure with filtration glomerular rate clearance less than 30ml / min.
* Diabetic neuropathy.
* Post menopause
* Intestinal malabsorption diseases .
* Type 2 diabetes with HbA1c > 8.5 %
* Systolic and diastolic blood pressure >140/90 mmHg.
* Triglycerides > 300 mg/dL.
* LDL cholesterol >160mg/dL.
* Systemic autoimmune diseases .
* Cirrhosis or liver failure .
* Subject infected with human immunodeficiency virus or acquired immunodeficiency syndrome .
* Diagnosis of cancer with active disease.
* Subject previously undergoing bariatric surgery.
* Pregnancy or lactation.
* Alcoholism and drug addiction.
* Subject who consume high fiber dietary supplements and / or omega 3 acids.
* Subject taking anorexic drugs.
* Subject under diet for weight loss implemented by a health professional.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Change in serum glucose levels | 94 days (plus or minus 4 days)
  Fasting, postprandial and post challenge oral test glucose and HbA1c
Variation in lipid profile | 94 days (plus or minus 4 days)
  Triglycerides, HDL-cholesterol, LDL-cholesterol and total cholesterol

SECONDARY OUTCOMES:
Modification in insulin resistance | 94 days (plus or minus 4 days)
  Serum insulin, homeostasis model assessment index
Change in systolic blood pressure | 94 days (plus or minus 4 days)
Change in diastolic blood pressure | 94 days (plus or minus 4 days)
Variation in body weight | 94 days (plus or minus 4 days)
Modification in waist circumference | 94 days (plus or minus 4 days)

CONTACTS AND LOCATIONS:
Overall Officials: Ana E Perez Verdin, MD, Principal Investigator
Locations (1):
- Instituto Mexicano Del Seguro Social Hospital de Especialidades, Centro Medico Nacional de Occidente Lic. Ignacio Garcia Tellez Unidad Medica de Alta Especialidad, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Result] Mohd Ali N, Yeap SK, Ho WY, Beh BK, Tan SW, Tan SG. The promising future of chia, Salvia hispanica L. J Biomed Biotechnol. 2012;2012:171956. doi: 10.1155/2012/171956. Epub 2012 Nov 21. PMID 23251075
- [Result] Ayerza R Jr, Coates W. Effect of dietary alpha-linolenic fatty acid derived from chia when fed as ground seed, whole seed and oil on lipid content and fatty acid composition of rat plasma. Ann Nutr Metab. 2007;51(1):27-34. doi: 10.1159/000100818. Epub 2007 Mar 14. PMID 17356263
- [Result] Chicco AG, D'Alessandro ME, Hein GJ, Oliva ME, Lombardo YB. Dietary chia seed (Salvia hispanica L.) rich in alpha-linolenic acid improves adiposity and normalises hypertriacylglycerolaemia and insulin resistance in dyslipaemic rats. Br J Nutr. 2009 Jan;101(1):41-50. doi: 10.1017/S000711450899053X. Epub 2008 May 20. PMID 18492301
- [Result] Rossi AS, Oliva ME, Ferreira MR, Chicco A, Lombardo YB. Dietary chia seed induced changes in hepatic transcription factors and their target lipogenic and oxidative enzyme activities in dyslipidaemic insulin-resistant rats. Br J Nutr. 2013 May;109(9):1617-27. doi: 10.1017/S0007114512003558. Epub 2012 Sep 5. PMID 22947172
- [Result] Oliva ME, Ferreira MR, Chicco A, Lombardo YB. Dietary Salba (Salvia hispanica L) seed rich in alpha-linolenic acid improves adipose tissue dysfunction and the altered skeletal muscle glucose and lipid metabolism in dyslipidemic insulin-resistant rats. Prostaglandins Leukot Essent Fatty Acids. 2013 Oct;89(5):279-89. doi: 10.1016/j.plefa.2013.09.010. Epub 2013 Sep 25. PMID 24120122
- [Result] Poudyal H, Panchal SK, Waanders J, Ward L, Brown L. Lipid redistribution by alpha-linolenic acid-rich chia seed inhibits stearoyl-CoA desaturase-1 and induces cardiac and hepatic protection in diet-induced obese rats. J Nutr Biochem. 2012 Feb;23(2):153-62. doi: 10.1016/j.jnutbio.2010.11.011. Epub 2011 Mar 22. PMID 21429727
- [Result] Vuksan V, Whitham D, Sievenpiper JL, Jenkins AL, Rogovik AL, Bazinet RP, Vidgen E, Hanna A. Supplementation of conventional therapy with the novel grain Salba (Salvia hispanica L.) improves major and emerging cardiovascular risk factors in type 2 diabetes: results of a randomized controlled trial. Diabetes Care. 2007 Nov;30(11):2804-10. doi: 10.2337/dc07-1144. Epub 2007 Aug 8. PMID 17686832
- [Result] Nieman DC, Cayea EJ, Austin MD, Henson DA, McAnulty SR, Jin F. Chia seed does not promote weight loss or alter disease risk factors in overweight adults. Nutr Res. 2009 Jun;29(6):414-8. doi: 10.1016/j.nutres.2009.05.011. PMID 19628108
- [Result] Jin F, Nieman DC, Sha W, Xie G, Qiu Y, Jia W. Supplementation of milled chia seeds increases plasma ALA and EPA in postmenopausal women. Plant Foods Hum Nutr. 2012 Jun;67(2):105-10. doi: 10.1007/s11130-012-0286-0. PMID 22538527
- [Result] Vuksan V, Jenkins AL, Dias AG, Lee AS, Jovanovski E, Rogovik AL, Hanna A. Reduction in postprandial glucose excursion and prolongation of satiety: possible explanation of the long-term effects of whole grain Salba (Salvia Hispanica L.). Eur J Clin Nutr. 2010 Apr;64(4):436-8. doi: 10.1038/ejcn.2009.159. Epub 2010 Jan 20. PMID 20087375
- [Result] Ho H, Lee AS, Jovanovski E, Jenkins AL, Desouza R, Vuksan V. Effect of whole and ground Salba seeds (Salvia Hispanica L.) on postprandial glycemia in healthy volunteers: a randomized controlled, dose-response trial. Eur J Clin Nutr. 2013 Jul;67(7):786-8. doi: 10.1038/ejcn.2013.103. Epub 2013 Jun 19. PMID 23778782
- [Result] Guevara-Cruz M, Tovar AR, Aguilar-Salinas CA, Medina-Vera I, Gil-Zenteno L, Hernandez-Viveros I, Lopez-Romero P, Ordaz-Nava G, Canizales-Quinteros S, Guillen Pineda LE, Torres N. A dietary pattern including nopal, chia seed, soy protein, and oat reduces serum triglycerides and glucose intolerance in patients with metabolic syndrome. J Nutr. 2012 Jan;142(1):64-9. doi: 10.3945/jn.111.147447. Epub 2011 Nov 16. PMID 22090467